CLINICAL TRIAL: NCT02530476
Title: Phase I/II, Study of Selective Inhibitor of Nuclear Export (SINE) Selinexor (KPT-330) + Sorafenib in Acute Myeloid Leukemia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Karyopharm Therapeutics Inc (Industry); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014-0975; NCI-2015-01523 (Other: NCI CTRP); P50CA100632 (NIH)
Record Dates: First submitted 2015-08-19; First posted 2015-08-21 (Estimated); Results first posted 2020-03-31 (Actual); Last update posted 2020-03-31 (Actual); Status verified 2020-03

CONDITIONS: Leukemia; Acute Myeloid Leukemia
Keywords: Leukemia; Acute myeloid leukemia; AML; Relapsed/Refractory; FLT3-ITD mutation; FLT3-mutated high-risk myelodysplastic syndrome; MDS; Chronic Myelomonocytic Leukemia; CMML; Selinexor; KPT-330; Sorafenib; Nexavar; BAY 43-9006; FLT3-inhibitor therapy
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid, Acute; Recurrence; Leukemia, Myelomonocytic, Chronic | interventions — selinexor; Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Phase I Group 1 Selinexor + Sorafenib (Experimental): Cohort includes those with FLT3-ITD and -D835 mutated participants with relapsed/refractory AML, including participants who may have been previously exposed to one or more FLT3-inhibitors.
  Phase I Starting Dose of Sorafenib: 400 mg by mouth twice daily for a 28 day cycle.
  Phase I Starting Dose of Selinexor: 80 mg by mouth twice weekly for a 28 day cycle.
  Interventions: Drug: Selinexor; Drug: Sorafenib
- Cohort 1 (FLT3-ITD inhibitor failure cohort) (Experimental): Cohort includes those with FLT3-ITD and -D835 mutated relapsed/refractory AML who have failed therapy with up to two prior salvage regimens.
  Phase II Starting Dose of Sorafenib: Maximum tolerated dose combination from Phase I.
  Phase II Starting Dose of Selinexor: Maximum tolerated dose from Phase I.
  Interventions: Drug: Selinexor; Drug: Sorafenib
- Cohort 2 (FLT3-ITD inhibitor naive cohort) (Experimental): Cohort includes those with FLT3-ITD and -D835 mutated relapsed/refractory AML who have failed therapy with up to two prior salvage regimens.
  Phase II Starting Dose of Sorafenib: Maximum tolerated dose combination from Phase I.
  Phase II Starting Dose of Selinexor: Maximum tolerated dose from Phase I.
  Interventions: Drug: Selinexor; Drug: Sorafenib
- Phase I Group 2 Selinexor + Sorafenib (Experimental): Cohort includes those with FLT3-ITD and -D835 mutated participants with relapsed/refractory AML, including participants who may have been previously exposed to one or more FLT3-inhibitors.
  Phase I Starting Dose of Sorafenib: 400 mg by mouth twice daily for a 28 day cycle.
  Phase I Starting Dose of Selinexor: 80 mg by mouth twice weekly for a 28 day cycle. Phase I Group 2 received Selinexor 80 mg by mouth twice weekly for a 28 day cycle.
  Interventions: Drug: Selinexor; Drug: Sorafenib

INTERVENTIONS:
Drug: Selinexor — Phase I Starting Dose of Selinexor: 80 mg by mouth twice weekly for a 28 day cycle.
  Phase II Starting Dose of Selinexor: Maximum tolerated dose from Phase I.
  Other Names: KPT-330
Drug: Sorafenib — Phase I Starting Dose of Sorafenib: 400 mg by mouth twice daily for a 28 day cycle.
  Phase II Starting Dose of Sorafenib: Maximum tolerated dose combination from Phase I.
  Other Names: Nexavar; BAY 43-9006

SUMMARY:
There are 2 parts to this study: Part 1 (dose escalation) and Part 2 (dose expansion).

The goal of Part 1 of this clinical research study is to find the highest tolerated dose of the combination of selinexor (KPT-330) and sorafenib (Nexavar) that can be given to patients with FLT3-ITD and -D835 mutated acute myeloid leukemia (AML) or FLT3-mutated high-risk myelodysplastic syndrome (MDS).

The goal of Part 2 of this study is to learn if the dose found in Part 1 can help to control the disease.

The safety of the drug combination will also be studied in both parts of this study.

This is an investigational study. Sorafenib is FDA approved and commercially available to treat hepatocellular cancer. Selinexor is not FDA approved or commercially available. It is currently being used for research purposes only. The combination of selinexor and sorafenib to treat FLT3-mutated AML and high-risk MDS is investigational.

The study doctor can explain how the study drugs are designed to work.

Up to 52 participants will take part in this study. All will be enrolled at MD Anderson.

DETAILED DESCRIPTION:
Study Groups:

If you are found to be eligible to take part in this study, you will be assigned to a study group based on when you join this study. Up to 3 groups of up to 6 participants will be enrolled in Part 1 of the study, and up to 40 participants will be enrolled in Part 2.

If you are enrolled in Part 1, the dose of selinexor and sorafenib you receive will depend on when you joined this study. The first group of participants will receive the starting dose combination level. If no intolerable side effects were seen, the next group will receive a higher dose of selinexor and sorafenib than Group 1. If intolerable side effects are seen, the next group may receive a lower dose level of selinexor and/or sorafenib. This will continue until the highest tolerable combination dose is found.

If you are enrolled in Part 2, you will receive selinexor and sorafenib at the highest tolerable combination dose or most effective combination dose found in Part 1.

Study Drug Administration:

Each study cycle is 28 days. However, the study cycles may be 3-12 weeks long, depending on if/how the disease responds to the treatment, how your bone marrow reacts to treatment, and what the doctor thinks is in your best interest.

You will take selinexor tablets by mouth 2 times each week (Monday/Wednesday or Tuesday/Thursday or Wednesday/Friday) for 3 weeks. You must take your dose of selinexor within 30 minutes after eating, with at least 4 ounces of fluids (either water, milk, juice, and so on). You must swallow the tablets whole. Do not crush them. If the powder comes into contact with your skin, you may have an increased chance of skin-related side effects.

You will take sorafenib by mouth 2 times a day, every day. Depending on how the disease responds to the study drugs, the number of days you receive the study drug may change. Your doctor will discuss this with you. You must take your dose of sorafenib at least 1 hour before or 1 hour after eating.

You will be given a drug diary and asked to write down what time you take the study drugs every day. You must bring in the study drug diary and any unused study drugs and bottles to each study visit.

Study Visits:

On Day 1 of Cycles 1-4 and then every 1-3 cycles after that:

* You will have a physical exam.
* You will have an EKG.

The study doctor will tell you how often you will have these tests after Cycle 4.

One time each week during Cycles 1-3, blood (about 1 tablespoon) will be drawn for routine tests. After Cycle 3, you will have this blood draw 1 time every 2-4 weeks. If the doctor thinks it is needed, blood may need to be drawn more often or more than 1 tablespoon of blood may need to be drawn.

After Cycle 1, you may be able to have these blood draws performed at a local lab or clinic that is closer to your home. The results of the testing will be sent to MD Anderson for review. The study doctor or study staff will discuss this option with you.

On Day 28 of Cycles 1 and 3 (+/- 7 days) and then every 1-3 cycles after that, you will have a bone marrow aspiration and/or biopsy to check the status of the disease.

Every 3 months (+/- 14 days), if you can become pregnant, blood (about 1-2 tablespoons) or urine will be collected for a pregnancy test.

If you stay on study for more than 6 months and you are not having side effects, you may have some of the above tests more or less often. The study doctor will discuss this with you.

Length of Study:

You may continue taking the study drugs for as long as the study doctor thinks it is in your best interest. You will no longer be able to take the study drugs if the disease gets worse, if intolerable side effects occur, or if you are unable to follow study directions.

Your participation on the study will be over after the follow-up visits.

End-of-Study Visit:

If you stop taking the study drugs before the end of Cycle 24:

* You will have a physical exam.
* Blood (about 2-3 tablespoons) will be drawn for routine tests.
* If the doctor thinks it is needed, you will have a bone marrow aspirate to check the status of the disease.

Follow-Up:

About 30 days (+/- 7) after your last dose of study drugs, you will have a physical exam. You may have this exam at MD Anderson or a local clinic near your home. If you have this exam at a local clinic, the results of the exam will be sent to MD Anderson for review.

If you cannot come to MD Anderson or a local clinic, you will be called by a member of the study staff and asked if you have had any side effects and/or started any new treatment(s). This call should last about 5 minutes.

Long-Term Follow-Up:

If the disease appears to get better and you are responding well to the study drug, you will return to MD Anderson every 3-6 months for up to 5 years after your last dose of study drugs for the study staff to check how you are doing.

If you cannot return to MD Anderson for these visits, you may be called by a member of the study staff. The call should last about 10 minutes.

ELIGIBILITY:
Inclusion Criteria:

1. FLT3-ITD and/or FLT3-D835 mutated patients 18 years of age or older with relapsed/ refractory AML (any number of relapses) including patients who may have been previously exposed to one or more FLT3-inhibitor therapies will be eligible for the phase I portion of this study.
2. Phase II FLT3-ITD and/or FLT3-D835 mutated relapsed/refractory patients: Patients should have a diagnosis of AML (de novo or transformed from hematologic malignancies). Patients with high-risk myelodysplastic syndrome (MDS) (defined as having >/= 10% blasts in the bone marrow) or patients with Chronic Myelomonocytic Leukemia (CMML) (having >/= 10% blasts in the bone marrow) may also be eligible after discussion with Principal Investigator (PI). The patients should have one of the following features: 1. Patients with AML should have failed any prior induction therapy or have relapsed after prior therapy. 2. Patients with high-risk MDS or high-risk CMML should have failed any prior therapy for the MDS or CMML. 3. Patients with MDS or CMML who received therapy for the MDS or CMML and progress to AML are eligible at the time of diagnosis of AML regardless any prior therapy for AML. The World Health Organization (WHO) classification will be used for AML.
3. Patients must be eligible for one of two cohorts: Cohort 1 (FLT3 and/or FLT3-D835 inhibitor failure cohort) in FLT3-ITD and/or FLT3-D835 mutated relapsed/refractory AML who have failed therapy with up to two prior salvage regimens (SCT or stem cell therapy for patients who previously underwent SCT/stem cell therapy in remission will not be considered a salvage regimen) and have previously been exposed at least one prior FLT3 inhibitor. Cohort 2 (FLT3 inhibitor naive cohort) in FLT3-ITD and/or FLT3-D835 mutated relapsed/refractory who have failed therapy with up to two prior salvage regimens (SCT or stem cell therapy for patients who previously underwent SCT/stem cell therapy in remission will not be considered a salvage regimen) with no prior exposure to any FLT3 inhibitor.
4. Age >/=18 years
5. Eastern Cooperative Oncology Group (ECOG) Performance Status </=2
6. Patients should have estimated life expectancy of >3 months at study entry
7. Adequate hepatic (serum total bilirubin </= 2.0 x upper limit normal (ULN) (or </= 3.0 x ULN if deemed to be elevated due to leukemia), alanine aminotransferase and/or aspartate transaminase </= 3.0 x ULN (or </= 5.0 x ULN if deemed to be elevated due to leukemia), and renal function (creatinine </= 2.0 mg/dL).
8. Patients must provide written informed consent.
9. In the absence of rapidly progressing disease, the interval from prior treatment to time of initiation of selinexor and sorafenib administration will be at least 2 weeks for cytotoxic agents or at least 5 half-lives for cytotoxic/noncytotoxic agents. The use of chemotherapeutic or anti-leukemic agents is not permitted during the study with the following exceptions: (1) intrathecal (IT) therapy for patients with controlled Central Nervous System (CNS) leukemia at the discretion of the PI and with the agreement of the Sponsor. Controlled CNS leukemia is defined by the absence of active clinical signs of CNS disease and no evidence of CNS leukemia on the most recent 2 simultaneous CSF evaluations. (2) Use of one dose of cytarabine (up to 2 g/m2) or hydroxyurea for patients with rapidly proliferative disease is allowed before the start of study therapy and for the first four weeks on therapy. These medications will be recorded in the case-report form.
10. Baseline ejection fraction must be >/= 40%.
11. Females must be surgically or biologically sterile or postmenopausal (amenorrheic for at least 12 months) or if of childbearing potential, must have a negative serum or urine pregnancy test within 72 hours before the start of the treatment.
12. Women of childbearing potential must agree to use an adequate method of contraception during the study and until 3 months after the last treatment. Males must be surgically or biologically sterile or agree to use an adequate method of contraception during the study until 3 months after the last treatment. Adequate methods of contraception include: Total abstinence when this is in line with the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception. Female sterilization (have had surgical bilateral oophorectomy with or without hysterectomy) or tubal ligation at least six weeks before taking study treatment. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment
13. (Continued from Criteria 12) Male sterilization (at least 6 months prior to screening). For female patients on the study, the vasectomized male partner should be the sole partner for that patient Combination of any of the two following (a+b or a+c or b+c) Use of oral, injected or implanted hormonal methods of contraception or other forms of hormonal contraception that have comparable efficacy (failure rate <1%), for example hormone vaginal ring or transdermal hormone contraception Placement of an intrauterine device (IUD) or intrauterine system (IUS) Barrier methods of contraception: Condom or Occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/ vaginal suppository
14. (Continued from Criteria 13) In case of use of oral contraception, women should have been stable on the same pill before taking study treatment. Note: Oral contraceptives are allowed but should be used in conjunction with a barrier method of contraception due to unknown effect of drug-drug interaction. Women are considered post-menopausal and not of child bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g. age appropriate, history of vasomotor symptoms) or have had surgical bilateral oophorectomy (with or without hysterectomy) or tubal ligation at least six weeks ago. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment is she considered not of child bearing potential.

Exclusion Criteria:

1. Patients with known allergy or hypersensitivity to selinexor, sorafenib or any of its components.
2. Subject has concurrent, uncontrolled medical condition, laboratory abnormality, or psychiatric illness, which could place him/her at unacceptable risk.
3. Patients who have had any major surgical procedure within 14 days of Day 1.
4. Patients currently receiving any other standard or investigational therapy for the treatment of AML.
5. Patients unwilling or unable to comply with the protocol.
6. Patients receiving concomitant treatment with strong CYP3A4 inhibitors, unless such drugs are considered critical for the well being of the patient and not adequate alternatives are available. Strong CYP3A4 inhibitors include the following medications: itraconazole, ketoconazole, miconazole, voriconazole; amprenavir, atazanavir, fosamprenavir, indinavir, nelfinavir, ritonavir; ciprofloxacin, clarithromycin, diclofenac, doxycycline, enoxacin, isoniazid, ketamine, nefazodone, nicardipine, propofol, quinidine, telithromycin.
7. Patients with any severe gastrointestinal or metabolic condition that could interfere with absorption of oral medications.
8. Patients who are in blast transformation of chronic myeloid leukemia (CML). Prior MDS or CMML is acceptable.
9. Patient has a concurrent active malignancy under treatment.
10. Unstable cardiovascular function: • Symptomatic ischemia, or • Uncontrolled clinically significant conduction abnormalities (i.e., ventricular tachycardia on antiarrhythmic agents are excluded; 1st degree atrioventricular (AV) block or asymptomatic left anterior fascicular block/right bundle branch block (LAFB/RBBB) will not be excluded), or • Congestive heart failure (CHF) New York Heart Association (NYHA) Class ≥ 3, or • Myocardial infarction (MI) within 3 months. • Left ventricular ejection fraction < 40 %. • Hypertension > 140 mm Hg systolic or > 90 mm Hg diastolic with or without antihypertensive therapy.
11. Uncontrolled infection at the time of enrollment. Infections controlled on concurrent anti-microbial agents are acceptable, and anti-microbial prophylaxis per institutional guidelines is acceptable.
12. Known active hepatitis B virus (HBV) or C virus (HCV) infection; or known to be positive for HCV ribonucleic acid (RNA) or HBsAg (HBV surface antigen).
13. Known human immunodeficiency virus (HIV) infection.
14. Female subjects who are pregnant or breastfeeding.
15. Acute promyelocytic leukemia.
16. Any medical condition, which in the investigator's opinion, could compromise the patient's safety.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2015-12-08 (Actual); Primary Completion 2019-04-08 (Actual); Study Completion 2019-04-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Naval Daver, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Zhang W, Ly C, Ishizawa J, Mu H, Ruvolo V, Shacham S, Daver N, Andreeff M. Combinatorial targeting of XPO1 and FLT3 exerts synergistic anti-leukemia effects through induction of differentiation and apoptosis in FLT3-mutated acute myeloid leukemias: from concept to clinical trial. Haematologica. 2018 Oct;103(10):1642-1653. doi: 10.3324/haematol.2017.185082. Epub 2018 May 17. PMID 29773601
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: December 2015 to July 2018
Groups:
- Phase I Group 1 Selinexor + Sorafenib: Cohort includes those with FLT3-ITD and -D835 mutated participants with relapsed/refractory AML, including participants who may have been previously exposed to one or more FLT3-inhibitors.
  Phase I Starting Dose of Sorafenib: 400 mg by mouth twice daily for a 28 day cycle.
  Phase I Starting Dose of Selinexor: 80 mg by mouth twice weekly for a 28 day cycle.
  Selinexor: Phase I Starting Dose of Selinexor: 80 mg by mouth twice weekly for a 28 day cycle.
  Phase II Starting Dose of Selinexor: Maximum tolerated dose from Phase I.
  Sorafenib: Phase I Starting Dose of Sorafenib: 400 mg by mouth twice daily for a 28 day cycle.
  Phase II Starting Dose of Sorafenib: Maximum tolerated dose combination from Phase I.
- Cohort 1 (FLT3-ITD Inhibitor Failure Cohort); Cohort 2 (FLT3-ITD Inhibitor Naive Cohort): Cohort includes those with FLT3-ITD and -D835 mutated relapsed/refractory AML who have failed therapy with up to two prior salvage regimens.
  Phase II Starting Dose of Sorafenib: Maximum tolerated dose combination from Phase I.
  Phase II Starting Dose of Selinexor: Maximum tolerated dose from Phase I.
  Selinexor: Phase I Starting Dose of Selinexor: 80 mg by mouth twice weekly for a 28 day cycle.
  Phase II Starting Dose of Selinexor: Maximum tolerated dose from Phase I.
  Sorafenib: Phase I Starting Dose of Sorafenib: 400 mg by mouth twice daily for a 28 day cycle.
  Phase II Starting Dose of Sorafenib: Maximum tolerated dose combination from Phase I.
Period: Overall Study
Arm/Group | Phase I Group 1 Selinexor + Sorafenib | Phase I Group 2 Selinexor + Sorafenib | Cohort 1 (FLT3-ITD Inhibitor Failure Cohort) | Cohort 2 (FLT3-ITD Inhibitor Naive Cohort)
Started | 4 | 3 | 7 | 3
Completed | 4 | 3 | 7 | 3
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase I Group 1 Selinexor + Sorafenib | Phase I Group 2 Selinexor + Sorafenib | Cohort 1 (FLT3-ITD Inhibitor Failure Cohort) | Cohort 2 (FLT3-ITD Inhibitor Naive Cohort) | Total
Number analyzed (Participants) | 4 | 3 | 7 | 3 | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 0 | 4 | 1 | 6
  >=65 years | 3 | 3 | 3 | 2 | 11
Age, Continuous [Median (Full Range); unit: years] | 78.5 [24 to 81] | 68 [68 to 74] | 63 [38 to 75] | 77 [31 to 79] | 68 [24 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 3 | 2 | 9
  Male | 3 | 0 | 4 | 1 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 2 | 2 | 1 | 5
  White | 4 | 0 | 4 | 1 | 9
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 4 | 3 | 6 | 3 | 16

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) of Selinexor With Sorafenib
Description: MTD defined as the highest dose level with </= 1 out of 6 patients experience a dose limiting toxicity (DLT) during the first 28 days of treatment.
Time Frame: 28 days
Population: The Outcome Measure of MTD was the objective of the Phase I Selinexor + Sorafenib cohort only. Data for MTD were not collected for patients on Cohorts 1 and 2.
Measure: Number; unit: Milligrams
Arm/Group | Phase I Group 1 Selinexor + Sorafenib | Phase I Group 2 Selinexor + Sorafenib | Cohort 1 (FLT3-ITD Inhibitor Failure Cohort) | Cohort 2 (FLT3-ITD Inhibitor Naive Cohort)
Number analyzed (Participants) | 4 | 3 | 0 | 0
Milligrams | 60 | 60 |  |

2. Primary Outcome: Composite CR (CRc) Rate Defined as CR (Complete Remission) + CRp (Complete Remission With Incomplete Platelet Recovery) + CRi (Complete Remission With Incomplete Count Recovery) Within 3 Months of Treatment Initiation
Description: CRc Response criteria modified from International Working Group for AML. Responders obtain a Composite Complete Remission Rate (CRc) with or without cytogenetic response, hematologic improvements, and morphologic leukemia-free state. CRc rate is defined as the confirmed remission rate of all complete and incomplete CRs (i.e., CR+ CRp + CRi).
  CR: bone marrow regenerating normal hematopoietic cells & morphologic leukemia-free state, & ANC > 1×10^9/L, platelet count ≥100×10^9/L, & normal marrow differential with <5% blasts, & red blood cell (RBC) and platelet transfusion independent, no evidence of extramedullary leukemia. CRp: CR except for incomplete platelet recovery (<100×10^9/L). CRi: Same criteria for CR except incomplete hematological recovery with residual neutropenia (ANC ≤ 1 × 109/L) with or without thrombocytopenia (platelet count <100×109/L). No need to be RBC or platelet transfusion independent (modification to Cheson criteria).
Time Frame: 84 days, assessed following first three cycles of therapy of Selinexor with Sorafenib
Population: Of the four participants in the Phase I Group 1 Selinexor + Sorafenib arm, one participant was not evaluable for response. Of the seven participants in cohort 1, one participant was not evaluable for response. Of the three participants in cohort 2, one participant was not evaluable for response.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I Group 1 Selinexor + Sorafenib | Phase I Group 2 Selinexor + Sorafenib | Cohort 1 (FLT3-ITD Inhibitor Failure Cohort) | Cohort 2 (FLT3-ITD Inhibitor Naive Cohort)
Number analyzed (Participants) | 3 | 3 | 6 | 2
Participants | 2 | 0 | 3 | 0

3. Secondary Outcome: Overall Survival
Description: Time from date of treatment start until date of death due to any cause or last Follow-up.
Time Frame: Up to 15 months, on average 5 months
Population: Overall Survival was not an objective outlined for participants in Phase I Group's 1 and 2, therefore overall survival was not done for these participants. Of the seven participants in cohort 1, one participant was not evaluable for response. Of the three participants in cohort 2, one participant was not evaluable for response.
Measure: Median (Full Range); unit: Months
Arm/Group | Phase I Group 1 Selinexor + Sorafenib | Phase I Group 2 Selinexor + Sorafenib | Cohort 1 (FLT3-ITD Inhibitor Failure Cohort) | Cohort 2 (FLT3-ITD Inhibitor Naive Cohort)
Number analyzed (Participants) | 0 | 0 | 6 | 2
Months |  |  | 3.5 [0.9 to 14] | 2.3 [0.8 to 5.5]

4. Secondary Outcome: Event Free Survival
Description: Time from date of treatment start until the date of first objective documentation of disease-relapse.
Time Frame: Up to 6 months
Population: Event Free Survival was not an objective outlined for participants in Phase I Group's 1 and 2, therefore overall survival was not done for these participants. Of the seven participants in cohort 1, one participant was not evaluable for response. Of the three participants in cohort 2, one participant was not evaluable for response.
Measure: Median (Full Range); unit: Months
Arm/Group | Phase I Group 1 Selinexor + Sorafenib | Phase I Group 2 Selinexor + Sorafenib | Cohort 1 (FLT3-ITD Inhibitor Failure Cohort) | Cohort 2 (FLT3-ITD Inhibitor Naive Cohort)
Number analyzed (Participants) | 0 | 0 | 6 | 2
Months |  |  | 1.8 [0.4 to 5.0] | 2.1 [0.7 to 2.1]

ADVERSE EVENTS:
Time Frame: 2 years, 7 months
Arm/Group | Phase I Group 1 Selinexor + Sorafenib | Phase I Group 2 Selinexor + Sorafenib | Cohort 1 (FLT3-ITD Inhibitor Failure Cohort) | Cohort 2 (FLT3-ITD Inhibitor Naive Cohort)
All-Cause Mortality (participants affected / at risk) | 1/4 | 0/3 | 2/7 | 2/3
Serious Adverse Events (participants affected / at risk) | 4/4 | 3/3 | 6/6 | 3/3
Other Adverse Events (participants affected / at risk) | 3/4 | 3/3 | 6/7 | 1/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I Group 1 Selinexor + Sorafenib (N=4) | Phase I Group 2 Selinexor + Sorafenib (N=3) | Cohort 1 (FLT3-ITD Inhibitor Failure Cohort) (N=6) | Cohort 2 (FLT3-ITD Inhibitor Naive Cohort) (N=3)
Acute Kidney Injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchopulmonary Hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Febrile Neutropenia (Infections and infestations) | 0 (0) | 0 (0) | 3 (5) | 1 (1)
Fever (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal Disorders Other (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Administration Site Conditions (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infections (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 2 (3)
Intracranial Hemorrhage (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Lower Gastrointestinal Hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lung Infection (Infections and infestations) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Muscle Weakness Lower Limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neck Pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neoplasms benign, malignant and Unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (3) | 1 (1) | 0 (0)
Thrombocytopenia (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Pulmonary Edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rectal Hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 1 (2) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I Group 1 Selinexor + Sorafenib (N=4) | Phase I Group 2 Selinexor + Sorafenib (N=3) | Cohort 1 (FLT3-ITD Inhibitor Failure Cohort) (N=7) | Cohort 2 (FLT3-ITD Inhibitor Naive Cohort) (N=3)
Acute Kidney Injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 3 (6) | 3 (4) | 3 (4) | 1 (1)
Cardiac Disorders (Cardiac disorders) | 2 (3) | 1 (1) | 0 (0) | 0 (0)
Confusion (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 2 (3) | 2 (3) | 3 (5) | 1 (3)
Fatigue (General disorders) | 3 (4) | 2 (4) | 3 (5) | 1 (1)
Hyperbilirubinemia (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 2 (2) | 1 (2) | 3 (5) | 1 (2)
Infection Other (Infections and infestations) | 1 (1) | 0 (0) | 2 (4) | 0 (0)
Nausea/Vomiting (Gastrointestinal disorders) | 3 (6) | 1 (1) | 3 (3) | 1 (1)
Weakness (Musculoskeletal and connective tissue disorders) | 3 (4) | 0 (0) | 2 (2) | 0 (0)
Weight Loss (Investigations) | 2 (2) | 2 (2) | 3 (4) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-07-14): https://cdn.clinicaltrials.gov/large-docs/76/NCT02530476/Prot_SAP_000.pdf